CLINICAL TRIAL: NCT07123454
Title: A Modular Phase I/II Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Efficacy of AZD4512 Monotherapy or in Combination With Other Anticancer Agent(s), in Participants With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma (B-NHL) (Lumi-NHL)
Brief Title: A Phase I/II Study of AZD4512 Monotherapy or in Combination With Anticancer Agents in Participants With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Acronym: Lumi-NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9890C00001
Record Dates: First submitted 2025-07-24; First posted 2025-08-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: AZD4512; Non-Hodgkin Lymphoma (NHL); Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Intervention Model Description: The study consists of individual modules each evaluating the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary efficacy of AZD4512 as monotherapy or in combination with other anticancer treatments in participants with R/R B-NHL
  - Module 1: AZD4512 Monotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Module 1: AZD4512 Monotherapy dose escalation + backfill (Experimental): In Mod 1, the efficacy and safety of AZD4512 will be evaluated in R/R B-NHL. Module 1 will consist of both dose escalation and Pharmacodynamic/safety backfills which may be used to support MTD and/or Optimal biological dose (OBD)
  Interventions: Drug: AZD4512

INTERVENTIONS:
Drug: AZD4512 — AZD4512 is an antibody-drug conjugate targeting cluster of differentiation 22 (CD22) that will be administered via IV infusion

SUMMARY:
This is a Phase I/II open-label, global multicenter study to evaluate the safety and efficacy of AZD4512 monotherapy or in combination with other anticancer agent(s), in participants with Relapsed/Refractory B-cell Non-Hodgkin Lymphoma (B-NHL).

DETAILED DESCRIPTION:
Study D9890C00001 (Lumi-NHL) is modular study designed to evaluate the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and efficacy of AZD4512 monotherapy or in combination with other anticancer agent(s), in participants with Relapsed/Refractory B-NHL. Module 1 aims to study AZD4512 monotherapy at in participants in R/R B-NHL who have been exposed to at least 2 prior lines of therapy.

Additional modules in specific B-NHL subtypes with AZD4512 as monotherapy or in combination with other anticancer agent(s) may be added in the future

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible patients must be adults (≥18 years)
* Documented diagnosis of B-cell non-Hodgkin lymphoma (B-NHL) as per World Health Organization (WHO) 2021 classification. In the dose escalation phase, any B-NHL subtype is allowed (excluding some subtypes), while the backfill phase restricts inclusion to defined subtypes: large B-cell lymphomas (as defined as Diffuse large B-cell lymphoma (DLBCL), Grade 3b Follicular lymphoma (FL), double/triple hit lymphomas, high-grade (B-cell lymphoma) BCL, primary mediastinal Large B-cell lymphoma (LBCL), and transformed indolent lymphoma), mantle cell lymphoma, and follicular lymphoma grades 1-3a.
* Patients must have relapsed or refractory disease after at least two prior lines of therapy and lack additional standard options with survival benefit:

A)LBCL patients must have progressed after both anti-CD20 and at least one systemic chemotherapy regimen, and have considered-or be ineligible for-CAR-T, T cell engager, and stem cell transplant modalities.

B) Mantle cell lymphoma (MCL) patients must have had anti-CD20 and Bruton's Tyrosine Kinase (BTK) inhibitor.

C)FL patients should have failed anti-CD20 with active disease requiring therapy.

Additional criteria include measurable disease by Lugano 2014, Eastern Cooperative Oncology Group (ECOG) performance status ≤2, and adequate organ and bone marrow function (as specified by blood counts, cardiac ejection fraction, renal and hepatic parameters, and coagulation indices).

Key Exclusion criteria

* Patients are excluded if they have a diagnosis of post-transplant lymphoproliferative disease, Richter's transformation, Burkitt's lymphoma, or chronic lymphocytic leukemia (CLL)/ Small lymphocytic lymphoma (SLL), or if they have active Central nervous system (CNS) involvement from their B-NHL. Exclusion also applies to those who have received Chimeric antigen receptor-T (CAR-T) or T cell engager therapies within 90 days prior to Cycle 1 Day 1 (C1D1), any investigational drug or other systemic anticancer therapies (except low-dose corticosteroids) within 21 days or 5 half-lives, and curative radiation within 14 days (localized palliative radiotherapy is allowed).
* Other exclusions include allogeneic Hematopoietic stem cell transplantation (HSCT) within 180 days (unless stable without active (graft-versus-host disease) GVHD for ≥2 months), autologous HSCT within 90 days (unless resolved toxicities), major surgery within 28 days, use of strong CYP3A4 inhibitors or (corrected QT interval - prolonging agents at C1, or other malignancies within two years. Patients with unresolved ≥ Grade 2 AEs from prior therapy (except specified tolerable conditions), serious uncontrolled medical conditions, active infection within 14 days, or history/suspicion of significant interstitial lung disease/pneumonitis are also excluded.
* Females who are pregnant or breastfeeding are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with dose-limiting toxicities (DLTs) | Up to 4 weeks
  To identify the maximum tolerated dose (MTD) and/or doses of AZD4512 for subsequent evaluation in participants with R/R B-NHL
Frequency, duration, severity of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) | From the first dose up to and including 30 (+7) days after the last dose of study treatment , but prior to subsequent cancer therapy
  To assess the safety and tolerability of AZD4512 in participants with R/R B-NHL
Frequency of SAEs/AEs leading to discontinuation of AZD4512 | From the first dose up to and including 30 (+7) days after the last dose of study treatment , but prior to subsequent cancer therapy
  To assess the safety and tolerability of AZD4512 in participants with R/R B-NHL
Number of participants with clinically significant alterations in vitals signs and abnormal laboratory parameters | From the first dose up to and including 30 (+7) days after the last dose of study treatment , but prior to subsequent cancer therapy
  To assess the safety and tolerability of AZD4512 in participants with R/R B-NHL

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR, according to Lugano classification 2024, to evaluate the preliminary efficacy of AZD4512 monotherapy in participants with R/R B-NHL.
Complete response (CR) rate | Up to 2 years
  CR rate, according to Lugano classification 2024, to evaluate the preliminary efficacy of AZD4512 monotherapy in participants with R/R B-NHL.
Duration of response (DoR) | Up to 2 years
  DoR, according to Lugano classification 2024, to evaluate the preliminary efficacy of AZD4512 monotherapy in participants with R/R B-NHL.
Progression-free survival (PFS) | Up to 2 years
  PFS, according to Lugano classification 2024, to evaluate the preliminary efficacy of AZD4512 monotherapy in participants with R/R B-NHL.
Overall survival (OS) | Up to 2 years
  OS, defined as the time from the date of first dose until date of death, to evaluate the preliminary efficacy of AZD4512 monotherapy in participants with R/R B-NHL.
Area Under plasma concentration-time Curve (AUC) of AZD4512, total antibody and total unconjugated warhead | Up to 2 years
  To characterize the AUC of AZD4512 as monotherapy in participants with R/R B-NHL
Observed plasma (peak) drug concentration (Cmax) of AZD4512, total antibody and total unconjugated warhead | Up to 2 years
  To characterize the Cmax of AZD4512 as monotherapy in participants with R/R B-NHL
Trough concentration (Ctrough) of AZD4512, total antibody and total unconjugated warhead | Up to 2 years
  To characterize the Ctrough of AZD4512 as monotherapy in participants with R/R B-NHL
Half life of AZD4512, total antibody and total unconjugated warhead | Up to 2 years
  To characterize the Half life of AZD4512 as monotherapy in participants with R/R B-NHL
Time to reach peak or maximum observed concentration (tmax) of AZD4512, total antibody and total unconjugated warhead | Up to 2 years
  To characterize the Tmax of AZD4512 as monotherapy in participants with R/R B-NHL
Total clearance of AZD4512, total antibody and total unconjugated warhead | Up to 2 years
  To characterize the Total clearance of AZD4512 as monotherapy in participants with R/R B-NHL
The number and percentage of participants who develop anti-drug antibodies (ADAs) | Up to 2 years
  To determine the immunogenicity of AZD4512 as monotherapy in participants with R/R B-NHL

CONTACTS AND LOCATIONS:
Locations (18):
- United States (6):
  - Research Site, Irvine, California
  - Research Site, Jacksonville, Florida
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Franklin, Tennessee
- Research Site, Melbourne, Australia
- China (2):
  - Research Site, Chengdu
  - Research Site, Guangzhou
- Italy (2):
  - Research Site, Bologna
  - Research Site, Milan
- Japan (2):
  - Research Site, Bunkyō City
  - Research Site, Kōtoku
- Research Site, Seoul, South Korea
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries and Associations (EFPIA) and the Pharmaceutical Research and Manufacturers of America (PhRMA) Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/